CLINICAL TRIAL: NCT00152815
Title: Non-alcoholic Fatty Liver Disease (NAFLD) in HIV: The Role of Nutritional Interventions
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough eligible patients available
Sponsor: Johane Allard (Other)
Collaborators: Ontario HIV Treatment Network (Network)
Responsible Party: Sponsor-Investigator, Johane Allard, Gastroenterologist, Professor of Medicine, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-0297-B; ROGB139
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: HIV Infections; Fatty Liver
Keywords: HIV; non-alcoholic fatty liver disease
MeSH Terms: conditions — HIV Infections; Fatty Liver; Non-alcoholic Fatty Liver Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin E (Experimental): alpha-tocoperol, capsules, 2 per day
  Interventions: Drug: antioxidant vitamin E; Behavioral: weight reduction and exercise

INTERVENTIONS:
Drug: antioxidant vitamin E — Vitamin E 800IU per day for 12 months
Behavioral: weight reduction and exercise — Patients will be asked to consume a self-selected, low fat, low-calorie diet of approximately 1200 kcal/d, which is consistent with American Heart Association guidelines for healthy weight reduction. Subjects will be provided with a videotape involving a structured 20 min aerobic exercise to be performed 3x/week.
  Other Names: This arm was removed from the study protocol, as the enrollment was slow and; a high drop-out rate was observed in the weigh-loss arm

SUMMARY:
The purpose of this study is to evaluate the effect of a one-year nutritional intervention with either betaine or vitamin E supplementation, or a weight reducing diet and exercise program on liver steatosis and steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Baseline liver biopsy with macrovesicular fatty degeneration with inflammation (lobular or portal), with or without Mallory bodies, hepatocyte damage, and/or fibrosis diagnostic of NAFLD
* Convincing evidence of negligible alcohol consumption (< 20 grams of ethanol per day) obtained from a detailed history, confirmed by at least one close relative
* If hyperlipidemia or diabetes, stable drug regimen required for the 6 months prior to and during the study
* Willingness to maintain stable weight and normal exercise program for the duration of the study, if randomized to vitamin E or betaine

Exclusion Criteria:

* Liver disease of other etiology diagnosed as per routine medical investigation (e.g., chronic viral hepatitis, auto-immune chronic hepatitis, primary biliary cirrhosis or genetic liver disease such as Wilson's disease, hemochromatosis, alpha-1 antitrypsin deficiency, or biliary obstruction)
* Complications of liver disease such as recurrent variceal bleeding, resistant ascites, spontaneous portosystemic encephalopathy, or bacterial peritonitis
* Concurrent medical illness contra-indicating a liver biopsy, history of unexplained bleeding, hemophilia or abnormal coagulation results as per routine laboratory work-up or other reason judged by the hepatologist to contra-indicate a percutaneous liver biopsy
* Medications known to precipitate steatohepatitis (corticosteroids, high dose estrogens, methotrexate, amiodarone, calcium channel blockers, spironolactone, sulfasalazine, naproxen, oxacillin or ampinovire) in the 6 months prior to entry
* Antioxidant vitamin supplementation, ursodeoxycholic acid, or any other experimental drug 6 months prior to study entry
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The change in grading of inflammation assessed by liver biopsy from month 0 to month 12 of the study | month 0 and month 12

SECONDARY OUTCOMES:
Liver histology for steatosis and fibrosis staging | month 0 and month 12
Liver immuno-histochemistry for adducts of MDA: a product of LP | month 0 and month 12
Alpha-smooth muscle actin (alpha-SMA): a marker of hepatic stellate cell activation | month 0 and month 12
Transforming growth factor (TGF-beta): a pro-fibrogenic cytokine involved in fibrogenesis | month 0 and month 12
Liver lipid peroxides and TNP-alpha | month 0, month 6 and month 12
  For oxidative stress and inflammation in the liver
Liver steatosis and volume will be assessed by ultrasound | month 0 and month 12
Liver enzymes and IR (HOMA and QUICKY) will also be measured | month 0, month 6 and month 12
Lipid peroxides, TNF-alpha, vitamin E and C in plasma | month 0, month 6 and month 12
  Parameters for oxidative stress and antioxidant capacity

CONTACTS AND LOCATIONS:
Overall Officials: Allard Johane, MD, FRCPC, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada